CLINICAL TRIAL: NCT06736717
Title: A Phase 1b/2 Trial of Onvansertib in Combination With NALIRIFOX for First Line Treatment of Advanced Pancreatic Cancer
Brief Title: Onvansertib in Combination With NALIRIFOX for First Line Treatment of Advanced Pancreatic Cancer
Acronym: PANCONVA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Cardiff Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00161071
Record Dates: First submitted 2024-11-20; First posted 2024-12-17 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — onvansertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Study Drug: Onvansertib:
  Orally daily on D1 - 5 of each 14-day cycle
  NALIRIFOX Intravenous D1 of each 14-day cycle
  Interventions: Drug: Onvansertib; Drug: NALIRIFOX

INTERVENTIONS:
Drug: Onvansertib — 20 or30mg flat dose - depending on results from safety lead-in. Administered concurrently with NALIRIFOX.
  Once daily on D1-5 of each 14-day cycle.
  Other Names: PCM-075; NMS-1286937
Drug: NALIRIFOX — Chemotherapy regimen of nanoliposomal irinotecan, oxaliplatin, fluorouracil [5-FU], and leucovorin.
  Intravenously on Day 1 of each 14-day cycle.

SUMMARY:
Pancreatic cancer is a deadly disease and will be the second leading cause of cancer related death behind lung cancer by 2030. Over 62,000 people are diagnosed each year in the United States with about 90% succumbing to the disease within 5 years. In the metastatic setting, NALIRIFOX, FOLFIRINOX and nab-paclitaxel-gemcitabine are standard treatment options in patients with good performance status (Eastern Cooperative Oncology Group [ECOG] 0/1). All three combinations have shown a survival advantage over previously standard gemcitabine-based therapy, with 11.1 months overall survival (OS) for NALIRIFOX/FOLFIRINOX and 8.7 months for nab-paclitaxel-gemcitabine versus 6.7 months for gemcitabine alone. There is an urgent need to improve treatment of patients with current and emerging therapeutic strategies.

KRAS is the most common oncogene mutated in pancreatic adenocarcinoma, and it is mutated in nearly all tumors. Mutant KRAS is essential for PDAC growth, where the constitutive activated RAS proteins contribute to tumorigenesis, treatment resistance, and metastases. Despite research and drug development efforts focused on KRAS, no effective RAS inhibitors have been approved for the treatment of pancreatic cancer with KRAS mutation. The poor prognosis of KRAS-mutated PDAC patients and the absence of KRAS-targeted therapies, highlight the urgency to develop novel therapies aimed at KRAS.

This study will investigate onvansertib (also known as PCM-075 and NMS-1286937) as the first PLK1-specific adenosine triphosphate competitive inhibitor administered by oral route to enter clinical trials with proven antitumor activity in different preclinical models.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant to understand this study, and participant willingness to sign a written informed consent. Remote consenting will be allowed on a case-by-case basis, but will not replace in-person visits for labs/physical, etc.
* Males and females age ≥ 18 years
* ECOG Performance Status 0 - 1
* Measurable disease by RECIST 1.1
* Histologically or cytologically confirmed adenocarcinoma of the exocrine pancreas
* Locally advanced unresectable or metastatic disease who are treatment naive
* No previous systemic therapy in the metastatic setting
* Participant must be willing to submit archival tissue if available and sufficient - otherwise fresh biopsy collection will be performed at screening UNLESS it is deemed medically unsafe for the participant. If participant does not have archival tissue and is not able to undergo a fresh biopsy at this time, enrollment will be per the principal investigator's discretion
* Adequate organ function, defined as follows:

  * Leukocytes (White Blood Cell [WBC]) > 3 K/UL
  * Absolute Neutrophil Count >1.5K/UL
  * Platelets >100K/UL
  * Hemoglobin ≥ 9 g/dL(level must be maintained without transfusions)
  * Calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault equation
  * Total bilirubin ≤ 1.5 x ULN
* If known Gilbert's syndrome then discuss with principal investigator. Email documentation of discussion and approval will be saved and documented for source.
* Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
* Women of child-bearing potential (WOCBP) and men with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception listed in Child-Bearing Potential/Pregnancy section.

Exclusion Criteria:

* Simultaneously enrolled in any therapeutic clinical trial
* Current or anticipating use of other anti-neoplastic or investigational agents while participating in this study
* Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
* Is pregnant or breastfeeding
* Has a known allergic reaction to any excipient contained in the study drug formulation
* Active Grade 3 (per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.027) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment.
* Patient has had major surgery within 4 weeks prior to enrollment
* Untreated or symptomatic brain metastasis
* Gastrointestinal (GI) disorder(s) that, in the opinion of the Investigator, would significantly impede the absorption of an oral agent (e.g., intestinal occlusion, active Crohn's disease, ulcerative colitis, extensive gastric and small intestine resection)
* Unable or unwilling to swallow study drug
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure (CHF) Class II or higher according to the New York Heart Association (NYHA) Functional Classification, unstable angina pectoris, clinically significant cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection
* Known active infection with HIV, with measurable viral titer, and/or active infection with hepatitis B or C (patients who have had a hepatitis B virus immunization are eligible)
* Known active infection with SARS-CoV-2 where symptoms are present
* Clinically significant ascites or pleural effusions
* Patients with a history of other malignancies except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix or prostate, or other solid tumors curatively treated with no evidence of disease for > 2 years
* Any active disease condition that would render the protocol treatment dangerous or impair the ability of the patient to receive study drug per PI discretion.
* Any condition (e.g., psychological, geographical, etc.) that does not permit compliance with the protocol
* Treatment with any of the drugs listed in section with title; Prohibited or Restricted Concomitant Medications at the time of study treatment initiation. Planned concomitant use of medications known to prolong the QT/QTc interval according to institutional guidelines. Use of strong CYP3A4 or CYP2C19 inhibitors or strong CYP3A4 inducers. Patients currently receiving these agents who can be switched to alternate therapy are not excluded. Inhibitors should be stopped at least 1 week prior to the first dose of protocol therapy and inducers should be stopped at least 2 weeks prior to initiation of protocol therapy
* QT interval: Fridericia's correction (QTcF) > 470 milliseconds.

  * A single ECG is sufficient. Triplicate may be done per PI discretion. If triplicate ECG completed, the QTcF should be calculated as the arithmetic mean of the QTcF on triplicate ECGs. In the case of potentially correctible causes of QT prolongation that are readily corrected (e.g., medications, hypokalemia), the triplicate ECG may be repeated once during Screening and that result may be used to determine eligibility
  * Presence of risk factors for torsade de pointes, including family history of Long QT Syndrome or uncorrected hypokalemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Approximately 2 years
  Imaging RECIST 1.1

SECONDARY OUTCOMES:
Adverse Events | 2 years
  The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.025
Anti-tumor activity by Disease Control Rate (DCR) | 8 weeks
  Calculated as the percentage of participants that achieve any of the following at 8 weeks: complete response, partial response, or stable disease, as defined by RECIST v1.1.
Anti-tumor activity by Duration of Response (DOR) | 2 years
  Calculated as the average length of time between response to treatment and disease progression, defined per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Progression Free Survival (PFS) | 2 years
  The duration of time from start of treatment until objective tumor progression or death, as determined by medical record imaging
Overall Survival (OS) | 2 years
  Duration of time from start of treatment to death, determined by medical record

CONTACTS AND LOCATIONS:
Overall Officials: Anup Kasi, MD, MPH, Principal Investigator — The University of Kansas Cancer Center
Locations (1):
- The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] U.S. Food and Drug Administration. Drug Development and Drug Interactions / Table of Substrates, Inhibitors and Inducers. URL: https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers
- [Background] Smith TJ, Bohlke K, Lyman GH, Carson KR, Crawford J, Cross SJ, Goldberg JM, Khatcheressian JL, Leighl NB, Perkins CL, Somlo G, Wade JL, Wozniak AJ, Armitage JO; American Society of Clinical Oncology. Recommendations for the Use of WBC Growth Factors: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol. 2015 Oct 1;33(28):3199-212. doi: 10.1200/JCO.2015.62.3488. Epub 2015 Jul 13. PMID 26169616
- [Background] Alembic Pharmaceuticals Inc. FLUOROURACIL - fluorouracil injection, solution. Package Insert Revised 10-2023
- [Background] Hospira. OXALIPLATIN injection, for intravenous use. Package Insert Revised 09-2023
- [Background] National Institute of Health/National Cancer Institute - Cancer Therapy Evaluation Program (CTEP). Common Terminology Criteria for Adverse Events (CTCAE). URL: https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm#ctc_60
- [Background] United States Food and Drug Administration. FDA approves irinotecan liposome for first-line treatment of metastatic pancreatic adenocarcinoma. 02-13-2024. URL: https://www.fda.gov/drugs/resources-information-approved-drugs/fda-approves-irinotecan-liposome-first-line-treatment-metastatic-pancreatic-adenocarcinoma
- [Background] Cardiff Oncology. Investigator's Brochure - Onvansertib (also known as PCM-075 and NMS-1286937) Edition 13 dated 09-19-2023
- [Background] Weichert W, Kristiansen G, Schmidt M, Gekeler V, Noske A, Niesporek S, Dietel M, Denkert C. Polo-like kinase 1 expression is a prognostic factor in human colon cancer. World J Gastroenterol. 2005 Sep 28;11(36):5644-50. doi: 10.3748/wjg.v11.i36.5644. PMID 16237758
- [Background] Weichert W, Kristiansen G, Winzer KJ, Schmidt M, Gekeler V, Noske A, Muller BM, Niesporek S, Dietel M, Denkert C. Polo-like kinase isoforms in breast cancer: expression patterns and prognostic implications. Virchows Arch. 2005 Apr;446(4):442-50. doi: 10.1007/s00428-005-1212-8. Epub 2005 Mar 23. PMID 15785925
- [Background] Luo J, Emanuele MJ, Li D, Creighton CJ, Schlabach MR, Westbrook TF, Wong KK, Elledge SJ. A genome-wide RNAi screen identifies multiple synthetic lethal interactions with the Ras oncogene. Cell. 2009 May 29;137(5):835-48. doi: 10.1016/j.cell.2009.05.006. PMID 19490893
- [Background] Lenz H-J, Kasi A, Mendelsohn L, et al. A phase 1b/2 trial of the PLK1 inhibitor onvansertib in combination with FOLFIRI-bev in 2L treatment of KRAS-mutated (mKRAS) metastatic colorectal carcinoma (mCRC). JCO. 2022.40.4 suppl.100. URL: https://ascopubs.org/doi/10.1200/JCO.2022.40.4_suppl.100
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Wainberg ZA, Melisi D, Macarulla T, Pazo Cid R, Chandana SR, De La Fouchardiere C, Dean A, Kiss I, Lee WJ, Goetze TO, Van Cutsem E, Paulson AS, Bekaii-Saab T, Pant S, Hubner RA, Xiao Z, Chen H, Benzaghou F, O'Reilly EM. NALIRIFOX versus nab-paclitaxel and gemcitabine in treatment-naive patients with metastatic pancreatic ductal adenocarcinoma (NAPOLI 3): a randomised, open-label, phase 3 trial. Lancet. 2023 Oct 7;402(10409):1272-1281. doi: 10.1016/S0140-6736(23)01366-1. Epub 2023 Sep 11. PMID 37708904
- [Background] Wang J, Hu K, Guo J, Cheng F, Lv J, Jiang W, Lu W, Liu J, Pang X, Liu M. Suppression of KRas-mutant cancer through the combined inhibition of KRAS with PLK1 and ROCK. Nat Commun. 2016 May 19;7:11363. doi: 10.1038/ncomms11363. PMID 27193833
- [Background] Degenhardt Y, Lampkin T. Targeting Polo-like kinase in cancer therapy. Clin Cancer Res. 2010 Jan 15;16(2):384-9. doi: 10.1158/1078-0432.CCR-09-1380. Epub 2010 Jan 12. PMID 20068088
- [Background] Knecht R, Elez R, Oechler M, Solbach C, von Ilberg C, Strebhardt K. Prognostic significance of polo-like kinase (PLK) expression in squamous cell carcinomas of the head and neck. Cancer Res. 1999 Jun 15;59(12):2794-7. PMID 10383133
- [Background] Waddell N, Pajic M, Patch AM, Chang DK, Kassahn KS, Bailey P, Johns AL, Miller D, Nones K, Quek K, Quinn MC, Robertson AJ, Fadlullah MZ, Bruxner TJ, Christ AN, Harliwong I, Idrisoglu S, Manning S, Nourse C, Nourbakhsh E, Wani S, Wilson PJ, Markham E, Cloonan N, Anderson MJ, Fink JL, Holmes O, Kazakoff SH, Leonard C, Newell F, Poudel B, Song S, Taylor D, Waddell N, Wood S, Xu Q, Wu J, Pinese M, Cowley MJ, Lee HC, Jones MD, Nagrial AM, Humphris J, Chantrill LA, Chin V, Steinmann AM, Mawson A, Humphrey ES, Colvin EK, Chou A, Scarlett CJ, Pinho AV, Giry-Laterriere M, Rooman I, Samra JS, Kench JG, Pettitt JA, Merrett ND, Toon C, Epari K, Nguyen NQ, Barbour A, Zeps N, Jamieson NB, Graham JS, Niclou SP, Bjerkvig R, Grutzmann R, Aust D, Hruban RH, Maitra A, Iacobuzio-Donahue CA, Wolfgang CL, Morgan RA, Lawlor RT, Corbo V, Bassi C, Falconi M, Zamboni G, Tortora G, Tempero MA; Australian Pancreatic Cancer Genome Initiative; Gill AJ, Eshleman JR, Pilarsky C, Scarpa A, Musgrove EA, Pearson JV, Biankin AV, Grimmond SM. Whole genomes redefine the mutational landscape of pancreatic cancer. Nature. 2015 Feb 26;518(7540):495-501. doi: 10.1038/nature14169. PMID 25719666
- [Background] Biankin AV, Waddell N, Kassahn KS, Gingras MC, Muthuswamy LB, Johns AL, Miller DK, Wilson PJ, Patch AM, Wu J, Chang DK, Cowley MJ, Gardiner BB, Song S, Harliwong I, Idrisoglu S, Nourse C, Nourbakhsh E, Manning S, Wani S, Gongora M, Pajic M, Scarlett CJ, Gill AJ, Pinho AV, Rooman I, Anderson M, Holmes O, Leonard C, Taylor D, Wood S, Xu Q, Nones K, Fink JL, Christ A, Bruxner T, Cloonan N, Kolle G, Newell F, Pinese M, Mead RS, Humphris JL, Kaplan W, Jones MD, Colvin EK, Nagrial AM, Humphrey ES, Chou A, Chin VT, Chantrill LA, Mawson A, Samra JS, Kench JG, Lovell JA, Daly RJ, Merrett ND, Toon C, Epari K, Nguyen NQ, Barbour A, Zeps N; Australian Pancreatic Cancer Genome Initiative; Kakkar N, Zhao F, Wu YQ, Wang M, Muzny DM, Fisher WE, Brunicardi FC, Hodges SE, Reid JG, Drummond J, Chang K, Han Y, Lewis LR, Dinh H, Buhay CJ, Beck T, Timms L, Sam M, Begley K, Brown A, Pai D, Panchal A, Buchner N, De Borja R, Denroche RE, Yung CK, Serra S, Onetto N, Mukhopadhyay D, Tsao MS, Shaw PA, Petersen GM, Gallinger S, Hruban RH, Maitra A, Iacobuzio-Donahue CA, Schulick RD, Wolfgang CL, Morgan RA, Lawlor RT, Capelli P, Corbo V, Scardoni M, Tortora G, Tempero MA, Mann KM, Jenkins NA, Perez-Mancera PA, Adams DJ, Largaespada DA, Wessels LF, Rust AG, Stein LD, Tuveson DA, Copeland NG, Musgrove EA, Scarpa A, Eshleman JR, Hudson TJ, Sutherland RL, Wheeler DA, Pearson JV, McPherson JD, Gibbs RA, Grimmond SM. Pancreatic cancer genomes reveal aberrations in axon guidance pathway genes. Nature. 2012 Nov 15;491(7424):399-405. doi: 10.1038/nature11547. Epub 2012 Oct 24. PMID 23103869
- [Background] Waters AM, Der CJ. KRAS: The Critical Driver and Therapeutic Target for Pancreatic Cancer. Cold Spring Harb Perspect Med. 2018 Sep 4;8(9):a031435. doi: 10.1101/cshperspect.a031435. PMID 29229669
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Hidalgo M. Pancreatic cancer. N Engl J Med. 2010 Apr 29;362(17):1605-17. doi: 10.1056/NEJMra0901557. No abstract available. PMID 20427809
- [Background] Ipsen Biopharmaceuticals, Inc. ONIVYDE® (irinotecan liposome injection) for intravenous use. Package Insert Revised 02-2023.
- See also: UpToDate. Causes of long QT syndrome — http://www.uptodate.com/contents/image?imageKey=CARD/57431